CLINICAL TRIAL: NCT02439229
Title: Decreased Femoral Bone Length by Fetal Ultrasound in Pregnant Women With Low Serum 25-hydroxyvitamin D: An Odense Child Cohort Study
Brief Title: The Vitamin D and Fetal Bone Length Study (VITFBL)
Status: Active, not recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Henrik Christesen, MD, PhD, Professor, Odense University Hospital
Other Study IDs: VITFBL
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Bone Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Vitamin D and fetal bone length study:

Vitamin D and its association to bone length in midterm pregnancy.

DETAILED DESCRIPTION:
Overall:

The Odense Child Cohort Study (OCC) is a population-based cohort study, comprising pregnant women recruited between January 1st 2010 and December 31st 2012. All women who were pregnant in the municipality of Odense during this time were eligible for participation, and 6,707 women were approached directly with recruitment material.

The study complied with the Helsinki declaration and was approved by the Regional Scientific Ethical Committee for Southern Denmark, no. S-20090130. All participants gave informed consent. From a population base of 6,707 pregnant women, 2,874 (42.9%) enrolled in the OCC up to December 31st, 2012. The children will be followed until 18 years of age.

Serum samples were taken in early pregnancy (GA 2-25 weeks), late pregnancy (GA 26-30 weeks), maternal serum and cord blood at birth, and from the children along with general examinations at ages 3 months, 1 year, 3 years.

Questionnaires were completed by the families in early pregnancy, late pregnancy, after birth, and at the times of clinical examination of the children.

Register data on health variables were further available from the Danish registries.

Objective:

The Vitamin D and bone length Study examines the relationship between the biomarker 25(OH)D in maternal serum and the length of the fetal femur and humerus bone at mid term pregnancy.

Method:

25(OH)D analysis: Serum was stored at -80º Celsius until analysis, which was performed by liquid chromatography mass spectrometry (LC-MS/MS). Triple deuterium marked 25(OH)vitamin D3 was added to serum samples as internal standard and deproteinized with ZnSO4 in methanol, centrifuged at 2750 g for 10 minutes, and 100 μl was injected on the TurboFlow column (Thermo Scientific) on the LC-MS/MS. The LC-MS/MS consisted of a Thermo Scientific TLX1 system connected to a Thermo Scientific Vantage TSQ. 25(OH)D2 and 25(OH)D3 were concentrated on a Thermo Scientific Cyclone P 50 x 1.0 mm column and back-flushed on the analytical column, Phenomenex Gemini C18 50 x 3.0 mm and eluted from the analytical column by a gradient. Mobile phases were A: 10 mM NH4Ac in water and B: 10 mM NH4Ac in methanol. Human serum was spiked with appropriate amounts of 25(OH)D2 and 25(OH)D3 in order to produce six point calibration curves (weighed 1/x2) and 3 levels of QC samples (low, mid, high). The method was calibrated against NIST standard 972.25 The C3 epimer of D3 was detected along with D3 and the two were not distinguishable from one another. Lowest detectable concentrations were 0.15 nM for both D2 and D3. Values of D2 and D3 were only considered if above 6.5 nM.

The Vitamin D and bone length study:

Vitamin D and bone length in mid term pregnancy.

- In 986 serum samples collected in early pregnancy, the levels of serum 25(OH)D were investigated by LC-MS/. Questionnaire and medical file information was used to determine the factors which were influential on 25(OH)D levels and bone length in mid term pregnancy by multiple linear regression.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and residing in the municipality of Odense during 2010-2012

Exclusion Criteria:

* Not residing in Odense, leaving the municipality

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The Odense Child Cohort Study (OCC) is a population-based cohort study, comprising pregnant women recruited between January 1st 2010 and December 31st 2012. All women who were pregnant in the municipality of Odense during this time were eligible for participation, and 6,707 women were approached directly with recruitment material.
  The study complied with the Helsinki declaration and was approved by the Regional Scientific Ethical Committee for Southern Denmark, no. S-20090130. All participants gave informed consent. From a population base of 6,70 pregnant women, 2,874 (42.9%) enrolled in the OCC up to December 31st, 2012. The children will be followed until 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 2874 (Actual)
Dates: Start 2010-01; Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Femur length | Outcome is assessed in gestational week 15+0 to 26+0.
  Size of femur bone length assessed by ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik T Christesen, MD, PhD, Principal Investigator — Project leader
Locations (1):
- HCA Research, Odense University Hospital, Odense, Denmark

REFERENCES:
- [Background] Christesen HT, Andersen LB. Reply to: 'vitamin D deficiency during pregnancy: confronting the issues'. Clin Endocrinol (Oxf). 2014 Jul;81(1):155-6. doi: 10.1111/cen.12328. Epub 2013 Oct 15. No abstract available. PMID 24102268
- [Background] Andersen LB, Abrahamsen B, Dalgard C, Kyhl HB, Beck-Nielsen SS, Frost-Nielsen M, Jorgensen JS, Barington T, Christesen HT. Parity and tanned white skin as novel predictors of vitamin D status in early pregnancy: a population-based cohort study. Clin Endocrinol (Oxf). 2013 Sep;79(3):333-41. doi: 10.1111/cen.12147. Epub 2013 Jul 2. PMID 23305099
- [Background] Galthen-Sorensen M, Andersen LB, Sperling L, Christesen HT. Maternal 25-hydroxyvitamin D level and fetal bone growth assessed by ultrasound: a systematic review. Ultrasound Obstet Gynecol. 2014 Dec;44(6):633-40. doi: 10.1002/uog.13431. PMID 24891235
- [Background] Christesen HT, Elvander C, Lamont RF, Jorgensen JS. The impact of vitamin D in pregnancy on extraskeletal health in children: a systematic review. Acta Obstet Gynecol Scand. 2012 Dec;91(12):1368-80. doi: 10.1111/aogs.12006. PMID 23210535
- [Background] Christesen HT, Falkenberg T, Lamont RF, Jorgensen JS. The impact of vitamin D on pregnancy: a systematic review. Acta Obstet Gynecol Scand. 2012 Dec;91(12):1357-67. doi: 10.1111/aogs.12000. Epub 2012 Oct 17. PMID 22974137
- [Background] Kyhl HB, Jensen TK, Barington T, Buhl S, Norberg LA, Jorgensen JS, Jensen DF, Christesen HT, Lamont RF, Husby S. The Odense Child Cohort: aims, design, and cohort profile. Paediatr Perinat Epidemiol. 2015 May;29(3):250-8. doi: 10.1111/ppe.12183. Epub 2015 Mar 10. PMID 25756293
- [Background] Lykkedegn S, Sorensen GL, Beck-Nielsen SS, Christesen HT. The impact of vitamin D on fetal and neonatal lung maturation. A systematic review. Am J Physiol Lung Cell Mol Physiol. 2015 Apr 1;308(7):L587-602. doi: 10.1152/ajplung.00117.2014. Epub 2015 Jan 16. PMID 25595644